CLINICAL TRIAL: NCT02969785
Title: An Intervention Program for the Trunk Neuromuscular Pattern and Postural Control in Athletes Chronic With Low Back Pain: A Feasibility and Clinical Trial Study
Brief Title: Postural Control and Trunk Neuromuscular Activation in Athletes With Chronic Low Back Pain
Acronym: PCMALBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Rubens Alexandre da Silva Jr, Professor, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rubens A. da Silva
Record Dates: First submitted 2016-11-11; First posted 2016-11-21 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Athletic Injury; Low Back Pain
Keywords: Postural control; Physiotherapy; Sports injuries; Low back pain; training
MeSH Terms: conditions — Athletic Injuries; Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1: exercises for lumbar stabilization (Experimental): Specific exercises for lumbar stabilization. The Group 1 (G1) will perform therapy with specific exercises for lumbar stabilization whith the Swiss ball as a therapeutic resource, including warming; stretching of hamstrings, paraspinals, trapezes; phasic perineal exercise; tonic perineal exercise; pelvic lumbar synergism; trunk mobility; mobility of the shoulder girdle; balance; and slow pelvic balance.
  Interventions: Other: G1: exercises for lumbar stabilization
- G2: back strengthening exercises (Active Comparator): Back strengthening exercises. The Group 2 (G2) will perform therapy including strengthning of back muscles on a Roman chair machine for flexion and extension of trunk with load progression from training volume for endurance and strength gains.
  Interventions: Other: G2: back strengthening exercises

INTERVENTIONS:
Other: G1: exercises for lumbar stabilization — Specific exercises for lumbar stabilization. The Group 1 (G1) will perform therapy with specific exercises for lumbar stabilization whith the Swiss ball as a therapeutic resource, including warming; stretching of hamstrings, paraspinals, trapezes; phasic perineal exercise; tonic perineal exercise; pelvic lumbar synergism; trunk mobility; mobility of the shoulder girdle; balance; and slow pelvic balance.
  Other Names: therapeutic exercises
  Arms: G1: exercises for lumbar stabilization
Other: G2: back strengthening exercises — Specific back exercises. The Group 2 (G2) will perform therapy including back strengthing exercise on a Roman chair machine to perform flexion and extension of trunk with load progressive training.
  Other Names: Back resistive training
  Arms: G2: back strengthening exercises

SUMMARY:
The relevance of this study is given by the feasibility to assess the effect of an intervention program based on the postural control and trunk neuromuscular activity, comparing two methods: stabilization exercises vs. back strengthening exercises, in athletes with low back pain. The main outcomes will be computed by electromyography measurement so that to assess the trunk neuromuscular activation pattern as well as by force platform parameters for determining of postural control. Clinical symptoms such as pain intensity, perception of disability and fear and avoidance will also be computed. This is the first study to compare two intervention methods using the main biological outcomes related to trunk neuromuscular function.

DETAILED DESCRIPTION:
For this study, a proposal of a 8-week intervention program will be carried out with lumbar stabilization exercises and back strengthening exercises, in 32 athletes with chronic low back, recruited by convenience and voluntaries from the community local and sports centers. Before intervention, all participantes will be evaluated by: electromoyography during back endurance and strength tests, balance performance, physical capacity, and by clinical outcomes such as pain, disability and psychological factors. All baseline testing and evaluation will be performed by a blinded evaluator to the study intervention. Afterwards, the participants will be randomized in two groups by a blinded evaluator (people not enroled to study): G1: exercises for lumbar stabilization; and G2: strengthening exercises. The intervention will follow 8 weeks, with 50 minutes of duration each session of therapy including measurement of blood pressure, heart rate and the Visual Analogue Scale (VAS) before and after each session, and the perception of exercise intensity monitored by Borg Scale. Within this proposal, the exercise sessions will performed twice a week. The intervention will follow the CONSORT recommendations for randomized controlled trials. The intervention will start in: G1 (n=16, motor control group), which will perform therapy with specific exercises for lumbar stabilization including the Swiss ball as therapeutic resource; while G2 (n=16, strength group) will perform back endurance progressive and resisted exercises on a Roman chair. The participants will not be blind to the study due to the characteristic of the exercises that often reflect to the improvement of the symptoms. In case of eventual losses, the intention-to-treat method will be used for the analyses. After the intervention, all groups will be invited to come back to the laboratory to proceed the same evaluation from baseline (trunk activation during exercises, balance, and clinical outcomes). For the analysis two-way ANOVA with repeated measures will be performed to compare the effects of the intervention (two groups) and times (baseline vs. end 8-weeks measurement) and the effects of interaction (Groups x Times). The size effect also will be computed to determine the rate of the changes observed.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain at least for three months, in a unique or multiple episodes.
* low back pain of unknown origin and mechanical nature.
* athletes must be train or play five times in a week.
* athletes must be participate in some official competition.

Exclusion Criteria:

* previous surgery (locomotor appareil).
* discal herniation diagnosis.
* nerve root entrapment.
* spondylolisis.
* spondylolisthesis;
* lumbar stenosis.
* hip cartilage damage.
* labral injury,
* piriformis syndrome.
* neurological disease.
* no current treatment in Physiotherapy or Pilates or Manual Therapy.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Eletromyography measurement | Change from baseline muscular activation at 8 weeks
  EMG estimates, Root Mean Square: RMS (in microvolts unit: uV) and Median Frequency: MF (in Hertz: Hz) will be computed to evaluate the back activation during strength maximal protocol and endurance dynamic test.

SECONDARY OUTCOMES:
Force platform measurement | Change from baseline muscular activation at 8 weeks
  Force platform measurement during balance performance using centre of pressure measures to assess balance performance.

OTHER OUTCOMES:
Visual Analogic Scale | Change from baseline muscular activation at 8 weeks
  Pain measurement using Short Version of Pain Questionnaire McGill (score 0 to 78; while higher score is determined by poor condition related to pain) and Visual Analogue Scale for pain intensity (score of 0 to 10 intensity; being 10 of poor score for VAS).
Disability questionnaire | Change from baseline muscular activation at 8 weeks
  Disability measurement using Oswestry questionnaire.
Fear-avoidance questionnaire | Change from baseline muscular activation at 8 weeks
  Fear-avoidance model measurement using Waddel questionnaire related to work and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens da Silva, PhD, Study Director — Laboratory of Functional Assessment and Human Motor Performance (LAFUP)
Locations (1):
- Laboratory of Functional Assessment and Human Motor Performance (LAFUP), Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Searle A, Spink M, Ho A, Chuter V. Exercise interventions for the treatment of chronic low back pain: a systematic review and meta-analysis of randomised controlled trials. Clin Rehabil. 2015 Dec;29(12):1155-67. doi: 10.1177/0269215515570379. Epub 2015 Feb 13. PMID 25681408
- [Background] Moon HJ, Choi KH, Kim DH, Kim HJ, Cho YK, Lee KH, Kim JH, Choi YJ. Effect of lumbar stabilization and dynamic lumbar strengthening exercises in patients with chronic low back pain. Ann Rehabil Med. 2013 Feb;37(1):110-7. doi: 10.5535/arm.2013.37.1.110. Epub 2013 Feb 28. PMID 23525973
- [Background] Cairns MC, Foster NE, Wright C. Randomized controlled trial of specific spinal stabilization exercises and conventional physiotherapy for recurrent low back pain. Spine (Phila Pa 1976). 2006 Sep 1;31(19):E670-81. doi: 10.1097/01.brs.0000232787.71938.5d. PMID 16946640
- [Background] McGill SM, Karpowicz A. Exercises for spine stabilization: motion/motor patterns, stability progressions, and clinical technique. Arch Phys Med Rehabil. 2009 Jan;90(1):118-26. doi: 10.1016/j.apmr.2008.06.026. PMID 19154838